CLINICAL TRIAL: NCT01948284
Title: A Randomized, Controlled Trial Comparing Maximal and Half-maximal Suction Pressure Applied During Water Exchange in Colonoscopy
Brief Title: Comparing Maximal and Half-maximal Suction Pressure Applied During Water Exchange in Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dalin Tzu Chi General Hospital (Other)
Collaborators: Felix Leung, MD, Sepulveda Ambulatory Care Center, VAGLAHS (Unknown)
Responsible Party: Principal Investigator, Yu-Hsi hsieh, Chief of Gastrointestinal Endoscopic Suite, Dalin Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DalinTzuChi-Hsieh-2013-2
Record Dates: First submitted 2013-09-17; First posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Minimally Sedated Patient Undergoing Colonoscopy
Keywords: cecal intubation time; water exchange; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- maximal suction pressure (Active Comparator): The pressure level of the suction unit (DF 601, Hanlien, Taipei, Taiwan) will be set at the maximal (-70 cm Hg).
  Interventions: Procedure: maximal pressure; Device: Suction Unit
- half-maximal pressure (Active Comparator): The pressure level of the suction unit will be set at the half-maximal (-35 cm Hg).
  Interventions: Procedure: half-maximal pressure; Device: Suction Unit

INTERVENTIONS:
Procedure: half-maximal pressure — the pressure level of the suction unit (DF 601, Hanlien, Taipei, Taiwan) will be set at the half-maximal (-35 cm Hg).
  Arms: half-maximal pressure
Procedure: maximal pressure — The pressure level of the suction unit (DF 601, Hanlien, Taipei, Taiwan) will be set at the maximal (-70 cm Hg).
  Arms: maximal suction pressure
Device: Suction Unit
  Other Names: suction unit (DF 601, Hanlien, Taipei, Taiwan)

SUMMARY:
This prospective, randomize, controlled trial will compared maximal to half-maximal suction pressure applied during water exchange in patients undergoing minimally sedated colonoscopy. We test the hypothesis that maximal suction pressure is more efficient and causes shorter insertion time.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing minimally sedated colonoscopy performed by YHH

Exclusion Criteria:

* known history of obstructive lesions of the colon,
* allergy to meperidine,
* massive ascites,
* past history of partial colectomy, or
* refusal to provide written informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
cecal intubation time | 30 minutes

SECONDARY OUTCOMES:
infused water amount | 30 minutes
aspirated water amount | 30 minutes
pain score | 30 minutes
suction marks on the mucosa | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Buddhist Dalin Tzu Chi General Hospital, Chiayi City, Taiwan, Taiwan

REFERENCES:
- [Background] Leung FW, Amato A, Ell C, Friedland S, Harker JO, Hsieh YH, Leung JW, Mann SK, Paggi S, Pohl J, Radaelli F, Ramirez FC, Siao-Salera R, Terruzzi V. Water-aided colonoscopy: a systematic review. Gastrointest Endosc. 2012 Sep;76(3):657-66. doi: 10.1016/j.gie.2012.04.467. PMID 22898423
- [Background] Leung J, Mann S, Siao-Salera R, Ransibrahmanakul K, Lim B, Canete W, Samson L, Gutierrez R, Leung FW. A randomized, controlled trial to confirm the beneficial effects of the water method on U.S. veterans undergoing colonoscopy with the option of on-demand sedation. Gastrointest Endosc. 2011 Jan;73(1):103-10. doi: 10.1016/j.gie.2010.09.020. PMID 21184876
- [Background] Leung JW, Mann SK, Siao-Salera R, Ransibrahmanakul K, Lim B, Cabrera H, Canete W, Barredo P, Gutierrez R, Leung FW. A randomized, controlled comparison of warm water infusion in lieu of air insufflation versus air insufflation for aiding colonoscopy insertion in sedated patients undergoing colorectal cancer screening and surveillance. Gastrointest Endosc. 2009 Sep;70(3):505-10. doi: 10.1016/j.gie.2008.12.253. Epub 2009 Jun 24. PMID 19555938
- [Background] Wasan SK, Schroy PC 3rd. Water-assisted unsedated colonoscopy: does the end justify the means? Gastrointest Endosc. 2009 Mar;69(3 Pt 1):551-3. doi: 10.1016/j.gie.2008.10.045. No abstract available. PMID 19231498